CLINICAL TRIAL: NCT04079218
Title: The Impact of HIV on Accelerated Aging in the Female Genital Tract: a Pilot Trial of Topical Estradiol to Improve the Vaginal Microbiome and Symptoms of Vaginal Atrophy in Menopausal Women With HIV
Brief Title: Accelerated Genital Tract Aging in HIV: Estradiol Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kerry Murphy (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Novo Nordisk A/S (Industry); Irma L and Abram S Croll Charitable Trust (Unknown)
Responsible Party: Sponsor-Investigator, Kerry Murphy, Assistant Professor, Department of Medicine (Infectious Diseases), Albert Einstein College of Medicine
Organization: Albert Einstein College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10529; 1K23AG062400-01A1 (NIH)
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: HIV Infection; Vaginal Atrophy; Menopause; Menopause Related Conditions; Aging; Premature Aging; Atrophic Vaginitis; Dysbiosis; Vaginitis
Keywords: HIV Infection; Vaginal Atrophy; Menopause; Vaginal Microbiome; Microbiome; Dysbiosis; Aging; Premature Aging; Atrophic Vaginitis
MeSH Terms: conditions — HIV Infections; Aging, Premature; Atrophic Vaginitis; Dysbiosis; Vaginitis | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive treatment with estradiol vaginal tablets or no treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Estradiol Vaginal Insert (Experimental): Using a pre-loaded single-use plastic applicator, participants will insert one 10 microgram estradiol tablet intravaginally daily for 2 weeks and then one tablet twice weekly for the remainder of the study for a total of 12 weeks.
  Interventions: Drug: Estradiol Vaginal Insert
- No treatment (No Intervention): No intervention

INTERVENTIONS:
Drug: Estradiol Vaginal Insert — Using a pre-loaded single-use plastic applicator, participants will insert one 10 microgram estradiol tablet intravaginally daily for 2 weeks and then one tablet twice weekly for the remainder of the study for a total of 12 weeks.
  Other Names: Vagifem®; Vagifem (estradiol vaginal tablet)
  Arms: Estradiol Vaginal Insert

SUMMARY:
During menopause, there is a decrease in a hormone estrogen, which leads to aging of the vagina. Vaginal aging includes changes in the type and amount of healthy bacteria in the vagina, inflammation and a breakdown of natural barriers that keep the vagina healthy and protected from infections. Some menopausal women develop a condition called vaginal atrophy, which causes vaginal dryness, irritation, pain with sex, and itching. We are testing whether an estradiol tablet placed inside the vagina will lead to fewer changes in the types of bacteria present in the vagina, improve vaginal atrophy symptoms and ultimately keep the vagina healthier for a longer. This is important for women with HIV as they are living longer, healthier, sexually active lives due to successful treatment with antiretrovirals.

DETAILED DESCRIPTION:
HIV may be associated with premature aging in the female genital tract including alterations in the vaginal microbiome and mucosal inflammation, which may increase risk for vaginal atrophy, urinary tract infections (UTI) and other genital tract infections. This study will determine whether use of vaginal estradiol for 12 weeks in menopausal women living with HIV with symptomatic vaginal atrophy will improve atrophy symptoms and the vaginal microbiome and reduce mucosal inflammation thereby improving vaginal health. This study will include 50 participants randomized to treatment with a vaginal estradiol insert or no therapy for 12 weeks and will have 4 study visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Females aged 45-70
* Menopause defined by having no menstrual periods for 12 consecutive months, confirmed with serum follicle-stimulating hormone (FSH) level >40 IU/ml and serum estradiol level <20 pg/ml
* Symptomatic vaginal atrophy defined as reporting at least once per week in the past 30 days, 1 or more of the following symptoms of moderate or severe intensity: Dryness, Itching, Irritation, Soreness or pain OR Pain associated with sexual activity at least once
* Evidence of atrophy on exam, including thin, pale and dry vaginal and vulvar surfaces
* Agrees not to use vaginal products other than vaginal estradiol tablet during the clinical trial

Exclusion Criteria:

* Current or previous history of breast cancer or estrogen dependent neoplasia
* Current or past thromboembolic disease (deep vein thrombosis or pulmonary embolism, not including thrombophlebitis)
* Current or previous history of myocardial infarction or stroke
* Known blood clotting disorders including Protein C, Protein S and antithrombin deficiency, Factor V Leiden or prothrombin mutations
* Known severe liver disease including cirrhosis or active Hepatitis B
* History of adverse reaction to vaginal estradiol
* Current unexplained or unevaluated abnormal genital bleeding
* Current or suspected pregnancy
* If < age 55, had a hysterectomy and has at least one ovary
* Pelvic or vaginal surgery in the prior 60 days
* Use of systemic reproductive hormones in the past 2 months
* Antibiotic use in the past 30 days
* Use of immunosuppressive medications in the prior 60 days including biologics, chemotherapeutics or post-transplant immunosuppressive medications
* Use of any vaginal or vulvar preparations 1 month prior to enrollment
* Current active vaginal infection (diagnosed by wet mount at Visit 1 or 2)
* Any serious disease or chronic condition that might interfere with study compliance
* Unwilling to agree to the provisions of the protocol

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry J Murphy, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication of the main study findings, external investigators may contact the Principal Investigator Dr. Kerry Murphy for de-identified datasets.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months after publication
Access Criteria: De-identified electronic datasets of published results will be made available to external investigators in a format in which subsequent statistical analyses can be performed.

REFERENCES:
- [Background] Murphy K, Keller MJ, Anastos K, Sinclair S, Devlin JC, Shi Q, Hoover DR, Starkman B, McGillick J, Mullis C, Minkoff H, Dominguez-Bello MG, Herold BC. Impact of reproductive aging on the vaginal microbiome and soluble immune mediators in women living with and at-risk for HIV infection. PLoS One. 2019 Apr 26;14(4):e0216049. doi: 10.1371/journal.pone.0216049. eCollection 2019. PMID 31026271
- [Background] Shen J, Song N, Williams CJ, Brown CJ, Yan Z, Xu C, Forney LJ. Effects of low dose estrogen therapy on the vaginal microbiomes of women with atrophic vaginitis. Sci Rep. 2016 Apr 22;6:24380. doi: 10.1038/srep24380. PMID 27103314
- [Background] Hummelen R, Macklaim JM, Bisanz JE, Hammond JA, McMillan A, Vongsa R, Koenig D, Gloor GB, Reid G. Vaginal microbiome and epithelial gene array in post-menopausal women with moderate to severe dryness. PLoS One. 2011;6(11):e26602. doi: 10.1371/journal.pone.0026602. Epub 2011 Nov 2. PMID 22073175
- [Background] Brotman RM, Shardell MD, Gajer P, Fadrosh D, Chang K, Silver MI, Viscidi RP, Burke AE, Ravel J, Gravitt PE. Association between the vaginal microbiota, menopause status, and signs of vulvovaginal atrophy. Menopause. 2018 Nov;25(11):1321-1330. doi: 10.1097/GME.0000000000001236. PMID 30358729
- [Background] Mitchell CM, Reed SD, Diem S, Larson JC, Newton KM, Ensrud KE, LaCroix AZ, Caan B, Guthrie KA. Efficacy of Vaginal Estradiol or Vaginal Moisturizer vs Placebo for Treating Postmenopausal Vulvovaginal Symptoms: A Randomized Clinical Trial. JAMA Intern Med. 2018 May 1;178(5):681-690. doi: 10.1001/jamainternmed.2018.0116. PMID 29554173

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 participants were consented and randomized into the study. Of these, 51 completed the trial. One participant in the non treatment arm and 8 participants in the estradiol arm did not complete the study. An additional 19 participants were screened but deemed ineligible for the study and not randomized. There were no HIV negative participants in the trial. Study documents refer to two related but separate studies: a trial for HIV+ participants and another study which includes HIV- participants.
Period: Overall Study
Arm/Group | Estradiol Vaginal Insert | No Treatment
Started | 33 | 27
Completed | 25 | 26
Not Completed | 8 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol Vaginal Insert | No Treatment | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (4.66) | 59.5 (4.92) | 59.4 (4.75)
Age, Customized [Count of Participants; unit: Participants] — Customized age ranges were collected and reported as described in the study protocol.
  Participants
    45-55 years old | 4 | 6 | 10
    56-70 years old | 21 | 20 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 20 | 40
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51
Plasma HIV-1 Viral Load [Count of Participants; unit: Participants] — Plasma HIV-1 Viral Load was assessed at baseline as a dichotomous variable. The number of participants who were determined to have "Detectable" vs "Undetectable" HIV-1 load was summarized by study arm. A viral load of <40 copies/ml was defined as undetectable. A viral > or = 40 copies/ml was defined as detectable.
  Participants
    Detectable | 5 | 5 | 10
    Undetectable | 20 | 21 | 41
Vaginal Cytokine and Chemokine Concentrations [Mean (Standard Deviation); unit: pg/mL] — Concentrations of vaginal cytokines and chemokines in cervicovaginal lavage (CVL) was determined. Upon assay, concentrations for the following cytokines and chemokines as individually expressed was reported in picograms per milliliter (pg/mL): IL-1A, Interleukin-8 (IL8); Interferon-gamma inducible protein 10 (IP-10); Monocyte Chemoattractant Protein-1 (MCP-1); and Secretory Leukocyte Protease Inhibitor (SLPI). Concentrations are summarized by study arm using basic descriptive statistics.
  pg/mL
    IL-1A | 1.88 (0.701) | 1.93 (0.669) | 1.91 (0.68)
    IL-8 | 2.58 (0.675) | 2.33 (1.06) | 2.45 (0.89)
    IP-10 | 2.24 (0.740) | 1.96 (0.848) | 2.10 (0.80)
    MCP-1 | 1.28 (0.753) | 1.12 (0.972) | 1.20 (0.87)
    SLPI | 4.42 (0.584) | 4.47 (0.722) | 4.45 (0.65)
Vaginal Symptom Index (VSI) [Mean (Standard Deviation); unit: score on a scale] — VSI was assessed at baseline. The VSI is a composite measure, calculated as the mean of 5 vaginal symptoms: dryness, itching, irritation, soreness, dyspareunia. Each symptom was given a score of 0-3 corresponding to either no symptoms, mild, moderate, or severe symptoms.
  score on a scale | 1.13 (0.64) | 1.04 (0.61) | 1.08 (0.62)
Vaginal Microbiome - Detectable Lactobacillus Crispatus (L. Crispatus) [Count of Participants; unit: Participants] — The number/percentage of participants with detectable concentrations of the protective Lactobacillus species, L. crispatus, as quantified by lllumina MiSeq sequencing, is summarized by study arm. Population: Data was not collected for 3 participants in the 'Estradiol' study arm and 1 participant in the 'No Treatment' study arm at Visit 2 (baseline).
  Participants
    number analyzed (Participants) | 22 | 25 | 47
    (all) | 5 | 7 | 12
Vaginal Microbiome - Detectable Bacterial Vaginosis-Associated Species [Count of Participants; unit: Participants] — The number/percentage of participants with detectable concentrations of the three most common Bacterial Vaginosis-associated species: Gardnerella vaginalis (G. vaginalis); Fannyhessea vaginae (F. vaginae); and Prevotella bivia (P. bivia), as quantified by lllumina MiSeq sequencing, is summarized by study arm. Population: Data was not collected for 3 participants in the 'Estradiol' study arm and 1 participant in the 'No Treatment' study arm at Visit 2 (baseline).
  Participants
    G. vaginalis: number analyzed (Participants) | 22 | 25 | 47
    G. vaginalis | 14 | 14 | 28
    F. vaginae: number analyzed (Participants) | 22 | 25 | 47
    F. vaginae | 11 | 12 | 23
    P. bivia: number analyzed (Participants) | 22 | 25 | 47
    P. bivia | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Most Bothersome Symptom (MBS) of Vaginal Atrophy
Description: Change in the severity of MBS of vaginal atrophy as reported during the baseline visit was assessed at 12 weeks (Visit 5). During the baseline visit, participants were asked to identify their MBS and assess the severity of the MBS on an ordinal scale of "None," "Mild," "Moderate," or "Severe." During the follow-up visit at 12 weeks participants were again asked to identify and assess the severity of their MBS. The degree of severity of the MBS reported at baseline was then compared to the severity of the MBS reported at 12 weeks and categorically summarized and reported as either "Severity Increased" "Severity Decreased" or "No change in Severity" for the given MBS. Participants whose MBS reported at baseline changed during the follow-up visit at 12 weeks were excluded from the analysis. Participants who did not report an MBS during the baseline visit were also excluded. Data for each possible type of MBS is summarized by study arm.
Time Frame: Between baseline (Visit 2) and 12 weeks (Visit 5)
Population: Participants whose MBS reported at baseline changed during the follow-up visit at 12 weeks and participants who did not report a MBS during the baseline visit were excluded. The overall number of participants analyzed has been updated to reflect this.
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 21 | 16
Participants
  Itching: number analyzed (Participants) | 8 | 6
  Itching: Severity Increased | 0 | 1
  Itching: Severity Decreased | 8 | 4
  Itching: No change in Severity | 0 | 1
  Dryness: number analyzed (Participants) | 10 | 10
  Dryness: Severity Increased | 0 | 1
  Dryness: Severity Decreased | 9 | 3
  Dryness: No change in Severity | 1 | 6
  Soreness: number analyzed (Participants) | 1 | 0
  Soreness: Severity Increased | 0 | 0
  Soreness: Severity Decreased | 1 | 0
  Soreness: No change in Severity | 0 | 0
  Irritation: number analyzed (Participants) | 0 | 0
  Irritation: Severity Increased | 0 | 0
  Irritation: Severity Decreased | 0 | 0
  Irritation: No change in Severity | 0 | 0
  Dyspareunia: number analyzed (Participants) | 2 | 0
  Dyspareunia: Severity Increased | 0 | 0
  Dyspareunia: Severity Decreased | 2 | 0
  Dyspareunia: No change in Severity | 0 | 0

2. Primary Outcome: Vaginal Microbiome - Relative Abundance of Lactobacillus Crispatus (L. Crispatus)
Description: The relative abundance of the protective Lactobacillus species, L. crispatus, as quantified by lllumina MiSeq sequencing will be calculated by dividing the total number of L crispatus sequences detected in a sample by the total number of sequences from all bacterial species detected in the same sample. This proportion will be expressed as a percentage. The change in relative abundance between baseline (visit 2) and 12 weeks (visit 5) will be summarized by study arm.
Time Frame: Between baseline (Visit 2) and 6 weeks and 12 weeks (Visit 5)
Population: Samples were not available for microbiome studies for 3 participants in the 'Estradiol' study arm and 1 participant in the 'No Treatment' study arm at both Visits 2 & 5 therefore there is no microbiome data available nor will there be in the future for these participants. Vaginal swabs were also collected at 6 weeks for all participants however due to lack of funding, sequencing was not performed therefore the data is not available nor will it be in the future.
Measure: Mean (Standard Deviation); unit: change in percentage of sequences
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 22 | 25
change in percentage of sequences | -1.37 (4.25) | -6.9 (25.14)

3. Primary Outcome: Vaginal Microbiome - Quantitative Determination of Protective Lactobacilli Species
Description: Changes in the vaginal microbiome, specifically the quantities of protective Lactobacilli species (L. crispatus, L. jensenii and L. gasseri) as measured by quantitative PCR (qPCR) will be determined. The three Lactobacilli species will be identified and quantified in colony forming units per milliliter of sample (CFU/mL). Changes in abundance from baseline will be summarized by study arm using basic descriptive statistics.
Time Frame: Between baseline (Visit 2) and 6 weeks and 12 weeks (Visit 5)
Population: Though cervicovaginal lavage samples were collected and utilized for other outcome measures reported including cytokine levels, etc, the portion of the cervicovaginal lavage that was collected for qPCR for the quantitative determination of protective Lactobacilli species was not utilized as we did not have sufficient funding to run qPCR. Therefore qPCR was not performed on any sample at any time point. qPCR data is not available nor will it be available in the future.
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Vaginal Microbiome - Relative Abundance of Bacterial Vaginosis Associated Species
Description: The relative abundance of bacterial vaginosis (BV) associated bacterial species as quantified by lllumina MiSeq sequencing, will be calculated by dividing the total number of the individual BV-associated species sequences in a sample by the total number of sequences from all bacterial species detected in the same sample. This proportion will be expressed as a percentage. The change in relative abundance between baseline (visit 2) and 12 weeks (visit 5) will be summarized by study arm for the 3 most common BV-associated species; Gardnerella vaginalis (G. vaginalis); Fannyhessea vaginae (F. vaginae); and Prevotella bivia (P. bivia)
Time Frame: Between baseline (Visit 2) and 6 weeks and 12 weeks (Visit 5)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change in percentage of sequences
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 22 | 25
change in percentage of sequences
  G. vaginalis | 3.15 (27.69) | -1.22 (17.03)
  F. vaginae | -5.17 (7.49) | -1.14 (8.72)
  P. bivia | -0.82 (1.79) | -1.09 (2.75)

5. Secondary Outcome: Vaginal Microbiome - Quantitative Determination of Bacterial Vaginosis Associated Species
Description: Changes in quantities of BV-associated species as measured by quantitative PCR (qPCR) will be determined. BV-associated species will be detected and quantified in colony forming units per milliliter of sample (CFU/mL). Changes in abundance from baseline for each detected species will be summarized by study arm using basic descriptive statistics.
Time Frame: Between baseline (Visit 2) and 6 weeks and 12 weeks (Visit 5)
Population: Though cervicovaginal lavage samples were collected and utilized for other outcome measures reported including cytokine levels, etc, the portion of the cervicovaginal lavage sample collected for qPCR for the quantitative determination of bacterial vaginosis associated species was not utilized as we did not have sufficient funding to run qPCR. Therefore qPCR was not performed on any sample at any time point. qPCR data for these species is not available nor will it be available in the future.
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Vaginal Cytokine and Chemokine Concentrations
Description: Change in concentrations from baseline of vaginal cytokines and chemokines in cervicovaginal lavage (CVL) was determined. Following assay, concentrations for the following cytokines and chemokines, as individually expressed, were reported in picograms per milliliter (pg/mL): IL-1A, Interleukin-8 (IL8); Interferon-gamma inducible protein 10 (IP-10); Monocyte Chemoattractant Protein-1 (MCP-1); and Secretory Leukocyte Protease Inhibitor (SLPI). Change in concentrations for the respective cytokines and chemokines from baseline are summarized by study arm using basic descriptive statistics.
Time Frame: Between baseline (Visit 2) and 6 weeks and 12 weeks (Visit 5)
Population: CVL was collected at 6 weeks however due to insufficient funding, levels of cytokines and chemokines were not run at this time point. Therefore the data is not available nor will it be in the future.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 25 | 26
pg/mL
  IL-1A | 0.17 (0.53) | -0.07 (0.14)
  IL-8 | -0.07 (0.28) | 0.11 (0.07)
  IP-10 | -0.04 (0.23) | 0.02 (0.06)
  MCP-1 | -0.13 (0.02) | 0.04 (0.21)
  SLPI | 0.18 (0.03) | -0.07 (0.00)

7. Other Pre Specified Outcome: HIV-1 RNA Levels in the Genital Tract
Description: HIV-1 RNA testing from cervicovaginal lavage fluid will be used to assess HIV-1 concentrations in the genital tract. Concentrations will be summarized by study arm and subsequently analyzed by multivariate linear regression.
  Cervicovaginal lavage (CVL) fluid was collected for other measures however due to insufficient funding, CVL HIV-1 viral loads were not run at any time point therefore the data is not available, nor will it be available in the future.
Time Frame: Baseline and 6 and 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Immunoglobulin (Ig)A and IgG Coated Bacteria
Description: Relative differences in levels of live IgA+IgG+ coated, live IgA+IgG- coated, live IgA-IgG-coated and dead bacteria will be summarized using basic descriptive statistics and subsequently analyzed by multivariate linear regression.
  Vaginal swabs were collected for quantification of subsets of IgA and IgG coated bacteria however due to insufficient funding, sequencing of these samples has not been performed and therefore data is not available. If we are able to secure additional funding, the sequencing may be performed in the future.
Time Frame: Baseline and 6 and 12 weeks
Reporting Status: Not Posted

9. Post Hoc Outcome: Change in Vaginal Symptom Index (VSI)
Description: Change in VSI was determined between Visit 2 and Visit 5. The VSI is a composite measure, calculated as the mean of 5 vaginal symptoms: dryness, itching, irritation, soreness, dyspareunia. Each symptom was given a score of 0-3 corresponding to either no symptoms, mild, moderate, or severe symptoms.
Time Frame: Between Baseline (Visit 2) and 12 weeks (Visit 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 25 | 26
score on a scale | -1.01 (0.65) | -0.38 (0.62)

10. Post Hoc Outcome: Vaginal Microbiome - Detectable Lactobacillus Crispatus (L. Crispatus)
Description: The number/percentage of participants with detectable concentrations of the protective Lactobacillus species, L. crispatus, as quantified by lllumina MiSeq sequencing, is summarized by study arm.
Time Frame: 12 weeks (Visit 5)
Population: Data was not collected for 3 participants in the 'Estradiol' study arm and 1 participant in the 'No Treatment' study arm at Visit 5 (12 weeks) therefore data is not and will not be available. Samples were collected at 6 weeks however due to insufficient finding, sequencing was not performed at the 6 week timepoint and therefore is not available and will not be available in the future.
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 22 | 25
Participants | 3 | 5

11. Post Hoc Outcome: Vaginal Microbiome - Detectable Bacterial Vaginosis-Associated Species
Description: The number/percentage of participants with detectable concentrations of the three most common Bacterial Vaginosis-associated species: Gardnerella vaginalis (G. vaginalis); Fannyhessea vaginae (F. vaginae); and Prevotella bivia (P. bivia), as quantified by lllumina MiSeq sequencing, is summarized by study arm.
Time Frame: 12 weeks (Visit 5)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 22 | 25
Participants
  G. vaginalis | 11 | 16
  F. vaginae | 11 | 11
  P. bivia | 8 | 9

12. Post Hoc Outcome: Change in Vaginal Microbiome - Detectable Lactobacillus Crispatus (L. Crispatus)
Description: Change from baseline in the percentage of participants with detectable concentrations of the protective Lactobacillus species, L. crispatus, as quantified by lllumina MiSeq sequencing, is summarized by study arm. The value was obtained by calculating the percentage difference in participants with a detectable level at baseline (Visit 2) when compared to 12 weeks (Visit 5).
Time Frame: Between baseline (Visit 2) and 6 weeks and 12 weeks (Visit 5)
Population: as for outcome 10
Measure: Number; unit: percentage change detectable sequences
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 22 | 25
percentage change detectable sequences | -9.1 | -8.0

13. Post Hoc Outcome: Change in Vaginal Microbiome - Detectable Bacterial Vaginosis-Associated Species
Description: Change from baseline in the percentage of participants with detectable concentrations of the three most common Bacterial Vaginosis-associated species: Gardnerella vaginalis (G. vaginalis); Fannyhessea vaginae (F. vaginae); and Prevotella bivia (P. bivia), as quantified by lllumina MiSeq sequencing, is summarized by study arm. Values were obtained for each species by calculating the percentage difference in participants with a detectable level at baseline (Visit 2) when compared to 12 weeks (Visit 5).
Time Frame: Between baseline (Visit 2) and 6 weeks and 12 weeks (Visit 5)
Population: as for outcome 10
Measure: Number; unit: percentage change detectable sequences
Arm/Group | Estradiol Vaginal Insert | No Treatment
Number analyzed (Participants) | 22 | 25
percentage change detectable sequences
  G. vaginalis | -13.6 | 8.0
  F. vaginae | 0 | -4.0
  P. bivia | -13.6 | -24.0

ADVERSE EVENTS:
Time Frame: Up to 13 weeks following randomization
Description: The Division of AIDS (DAIDS) Female Genital Grading Table for Use in Microbicide Studies will be the primary tool for grading adverse events (https://rsc.niaid.nih.gov/sites/default/files/addendum-1-female-genitalgrading-table-v1-nov-2007.pdf.)
Arm/Group | Estradiol Vaginal Insert | No Treatment
All-Cause Mortality (participants affected / at risk) | 1/33 | 0/27
Serious Adverse Events (participants affected / at risk) | 4/33 | 2/27
Other Adverse Events (participants affected / at risk) | 20/33 | 10/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Vaginal Insert (N=33) | No Treatment (N=27)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Verbatim Term: Blood Sugar dropped. Patient was hospitalized. Grade 4
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Secondary to drug use. Determined by autopsy. Patient expired.
Hospitalization for Gastrointestinal Bleed (GIB) (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 4
Fractured Right Distal Fibula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Grade 3
Liver Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hospitalization for Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) — Admit for pulmonary edema and hypertensive emergency in setting of end stage renal disease and known underlying cardiac disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol Vaginal Insert (N=33) | No Treatment (N=27)
Pigmentation loss (Reproductive system and breast disorders) | 1 | 0 — Verbatim Term. Pigmentation loss of bilateral internal labia/complete vulvar area. Grade 3
Hemoglobin Decreased (Blood and lymphatic system disorders) | 1 | 2 — Verbatim Term: Hemoglobin levels 9.8 g/dL (chronic anemia), 10.0 g/dL and 10.3 g/dL. All Grade 1
Leg weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin Pain (Renal and urinary disorders) | 1 | 0 — Worsening of chronic condition. Secondary to non-obstructing kidney stone and myomatous uterus. Grade 1
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 1 — Both Grade 1
Urinary Frequency (Renal and urinary disorders) | 1 | 0 — Verbatim Term: More frequent urination at night. Grade 1
Brown (Vaginal) Discharge (Reproductive system and breast disorders) | 2 | 0 — Both Grade 1
Vaginal Cramping (Reproductive system and breast disorders) | 1 | 0 — Grade 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 — Grade 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 | 0 — Pruritic rash on left forearm. Grade 1
Edema Limbs (General disorders) | 1 | 1 — Verbatim Term: Lower extremity edema. Grade 1; Edema to medial/lateral foot after surgery. Grade 2
Vulvar Erythema (Reproductive system and breast disorders) | 0 | 1 — Bilateral. Grade 2
Trichomonas (Infections and infestations) | 1 | 1 — Grade 2
Yeast Infection (Infections and infestations) | 1 | 1 — Both Grade 1
Healing Biopsy Sites (Injury, poisoning and procedural complications) | 1 | 0 — Grade 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 — Grade 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 — One Grade 1 and one Grade 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 — Grade 1
Bacterial Vaginosis (Infections and infestations) | 1 | 1 — Grade 2
Constipation (Gastrointestinal disorders) | 1 | 0 — Secondary to GIB
Dark Stools (Gastrointestinal disorders) | 1 | 0 — Secondary to GIB
Hemoglobin decreased 8.7 (Blood and lymphatic system disorders) | 1 | 0 — Hemoglobin decreased from 10.1 to 8.7 in setting of heavy nose bleeds, grade 2
Epigastric pain (Gastrointestinal disorders) | 1 | 0 — ED visit for epigastric pain, symptoms treated and sent home. Grade 2
Headache (Nervous system disorders) | 1 | 0 — Seen in ED for worsening migraines, treated and sent home from ED. Grade 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — See in ED for bronchitis symptoms, treated and send home from ED. Grade 2
Chest pain (Gastrointestinal disorders) | 0 | 1 — Seen in ED for chest pain, attributed to acid reflux, treated and send home from ED. Grade 2
Diarrhea and abdominal cramping (Gastrointestinal disorders) | 1 | 0 — In setting of new medications including metformin and jardiance as well as a viral illness. Grade 2
Tooth extraction (Surgical and medical procedures) | 1 | 0 — Tooth extraction under local anesthesia, grade 1
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Sinus infection treated with antibiotics. Grade 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — Seen in ED for COPD exacerbation, treated and send home from ED. Grade 2; Hospitalized for COPD exacerbation. Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT04079218/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT04079218/ICF_001.pdf